CLINICAL TRIAL: NCT00547677
Title: A Phase I Trial of Stereotactic Radiosurgery for Patients With Hepatic Metastases (SBRT Liver)
Brief Title: Stereotactic Radiosurgery for Patients With Hepatic Metastases.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000571611; SCCC-062004-005
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: liver metastases; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: stereotactic radiosurgery

SUMMARY:
RATIONALE: Stereotactic radiosurgery may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

PURPOSE: This phase I trial is studying the side effects and best dose of stereotactic radiosurgery in treating patients with liver metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated dose of fractionated stereotactic radiosurgery in patients with hepatic metastases.
* To determine the dose-limiting toxicity of stereotactic radiosurgery in these patients.
* To assess the tumor response in these patients.

OUTLINE: This is a multicenter study.

Patients receive 3-5 fractions of stereotactic radiosurgery over 14 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 9-13 patients receive escalating doses of stereotactic radiosurgery until 60 Gy is reached or the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which > 33% of patients experience dose-limiting toxicity.

After completion of study therapy, patients are followed at 6 weeks, every 3 months for 1 year, every 6 months for 2 years, and then annually for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary cancer

  * Stage IV primary disease with up to five liver metastases that are visualized on CT scan, MRI of the abdomen, or positron-emission tomography

    * No liver metastases secondary to germ cell tumor or hematologic malignancy
    * Other sites of metastases allowed
* No malignant ascites
* The cumulative total dose of radiotherapy to ≥ 2/3 of the liver and surrounding normal tissues, including the esophagus, stomach, and small bowel, must be ≤ 15 Gy
* Percutaneous or laparoscopic biopsy of the metastasis and placement of 3-5 fiducials required if undergoing Cyberknife for treatment delivery

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 3 months
* Albumin ≥ 3 g/dL
* Alkaline phosphatase < 1.5 times upper limit of normal (ULN)
* AST and ALT < 1.5 times ULN
* Total bilirubin < 1.5 times ULN
* Prothrombin time < 1.5 times ULN
* Hemoglobin > 10 g/dL
* Platelet count > 100,000/mm³
* ANC > 1,000/mm³
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of diagnosed inflammatory bowel disease, such as ulcerative colitis or Crohn's disease
* No active peptic ulcer disease
* No hepato-renal syndrome

PRIOR CONCURRENT THERAPY:

* Prior systemic therapy allowed provided complete blood cell counts have recovered
* No other concurrent antineoplastic treatment

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of stereotactic radiosurgery as assessed by NCI CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Timmerman, MD, Study Chair — Simmons Cancer Center
Locations (2):
- United States (2):
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas